CLINICAL TRIAL: NCT03981692
Title: The Effect of Two Different Dual Task Balance Trainings on Balance and Gait in Older Adults
Brief Title: The Effect of Two Different Dual Task Balance Trainings in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2019.181
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Dual Task Exercises in Elderly People
Keywords: Elderly; Balance; Gait speed; Cognitive; Dual task

STUDY DESIGN:
Intervention Model Description: In the study; sit-up, stand on one leg (eye open-closed), standing 30 sec stop (eye open closed stop), 10 m walk backward, sitting on top of the ball (eye open-closed), transfer of weight on the top-left, walking in a straight line, 30 sec. stop on soft ground (eye open-close), balance training which does not force their efforts will be given in two groups.
  Group 1: Integrated Dual Task Training Group performed balance and cognitive tasks simultaneously.
  Group 2: Consecutive Dual Task Training Group performed balance and cognitive tasks sequentially.
  The cognitive tasks; They were expected to find the letters Z in the mixed letters, search for the five words you read on the previous page, find the similarities between the concepts, find the letter in the given tables, derive the fruit names starting with the letter, count the days of the week, etc. Attention, memory and arithmetic training will be given the ability to run.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consecutive Dual Task Training (Active Comparator): Sit-up, stand on one leg (eye open-closed), standing 30 sec stop (eye open closed stop), 10 m walk backward, sitting on top of the ball (eye open-closed), transfer of weight on the top-left, walking in straight line, 30 sec. stop on soft ground (eye open-close), balance training which does not force their efforts will be given to the group. Immediately after these trainings, they should expected to find the letters Z in the mixed letters, search for the five words you read on the previous page, find the similarities between the concepts, find the letter in the given tables, derive the fruit names starting with the letter, count the days of the week etc. Attention, memory and arithmetic training will be given the ability to run.
  Interventions: Other: Consecutive dual task
- Integrated Dual Task Training (Active Comparator): Sit-up, stand on one leg (eye open-closed), standing 30 sec stop (eye open closed stop), 10 m walk backward, sitting on top of the ball (eye open-closed), transfer of weight on the top-left, walking in straight line, 30 sec. stop on soft ground (eye open-close), balance training which does not force their efforts will be given to the group. They will be done similar cognitive activities during with this simple balance trainings.
  Interventions: Other: Integrated dual task

INTERVENTIONS:
Other: Consecutive dual task — 8 weeks and 2 days per week, one session 45 min. Consecutive dual task creates the idea that it may provide more workable work without creating stress while doing secondary task during dual task.
  Arms: Consecutive Dual Task Training
Other: Integrated dual task — 8 weeks and 2 days per week, one session 45 min. Integrated dual task is a proven mode of work that has positive effects on geriatrics
  Arms: Integrated Dual Task Training

SUMMARY:
The aim of our study is to investigate the effect of integrated and consecutive dual-task exercise trainings in elderly people on the balance, fear of falling and gait performance.

DETAILED DESCRIPTION:
For the purpose, the number of 42 participants reached by the power analysis method was determined as 60 people considering the possible separations. 60 participants will be included in the study. Participants should not have any orthopedic, neurological and cognitive disabilities and the Montreal Cognitive Assessment (MOCA) scale score should be 21 or higher. Participants will be divided into two groups as random consecutive and integrated dual activity groups.

In the study sit-up, stand on one leg (eye open-closed), standing 30 sec stop (eye open closed stop), 10 m walk backward, sitting on top of the ball (eye open-closed), transfer of weight on the top-left, walking in straight line, 30 sec. stop on soft ground (eye open-close), balance training which does not force their efforts will be given in two groups.

For the sequential dual activity group, immediately after these trainings, you should expected to find the letters Z in the mixed letters, search for the five words you read on the previous page, find the similarities between the concepts, find the letter in the given tables, derive the fruit names starting with the letter, count the days of the week etc. Attention, memory and arithmetic training will be given the ability to run. For the integrated dual activity group will be given similar cognitive tasks during simple balance training.

The training program will be prolonged 8 weeks and 2 days per week for both groups.

The assessment tests was performed before and after the program. Primer Outcome Measure: Berg Balance Scale, Timed Up and Go Test (Standart-Cognitive), 10m Walking Speed Test (under single and dual task conditions).

Although there are many studies to increase and measure the balance and physical capacity of elderly people in the literature, there is no study using consecutive exercises and comparing the benefits of consecutive and integrated cognitive dual task training.

A major cause of morbidity and mortality is a fall injury in the elderly. Therefore, preventing falls in elderly people and increasing the ability to balance is an important public health priority.

Our study aims to benefit the public health, the reduction of health expenses of our country, the physiotherapists working with elderly people and the literature.

ELIGIBILITY:
Inclusion Criteria:

* Accepts to start routine exercise programs under the supervision of the medical team,
* Over age 65,
* Does not have orthopedic problems that may prevent him from exercising,
* The MOCA score is 21 or higher,
* Participants who have no other neurological problems that may cause loss of balance will be taken.

Exclusion Criteria:

* Having orthopedic problems that prevent him from exercising,
* Being under the MOCA score 21,
* To have any neurological problem that will affect the balance,
* Not wanting to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | 15 minutes
  The Berg Balance Scale (or BBS) is a widely used clinical test of a person's static and dynamic balance abilities, named after Katherine Berg, one of the developers. For functional balance tests, the BBS is generally considered to be the gold standard.
  The test takes 15-20 minutes and comprises a set of 14 simple balance related tasks, ranging from standing up from a sitting position, to standing on one foot. The degree of success in achieving each task is given a score of zero (unable) to four (independent), and the final measure is the sum of all of the scores.
  Minimum score is 0 while maximum score is 56. The classification; 0-20 scores - wheelchair user, 21-44 scores - walking with assistance 45-56 scores - independent.
  The test was performed at baseline and after Intervention (8 weeks)

SECONDARY OUTCOMES:
Timed Up and Go test (TUGST) | 5 minutes
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Description of the Instrument. Patients are timed (in seconds) when performing the TUG-3 conditions 1. TUG alone-from sitting in a chair, stand up, walk 3 meters, turn around, walk back, and sit down.. 2. TUG Cognitive-complete the task while counting backwards from a randomly selected number between 20 and 100.
  The test was performed at baseline and after Intervention (8 weeks)
Timed Up and Go test Cognitive (TUGCOG) | 5 minutes
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Description of the Instrument. Patients are timed (in seconds) when performing the TUG-3 conditions 1. TUG alone-from sitting in a chair, stand up, walk 3 meters, turn around, walk back, and sit down.. 2. TUG Cognitive-complete the task while counting backwards from a randomly selected number between 20 and 100.
  When a cognitive task is added while performing the test, it is called Timed Up and Go Cognitive.
  The test was performed at baseline and after Intervention (8 weeks)
10 Meters Walking Test Under Dual Task Condition (10MWTDT) | 5 minutes
  The standard 10 m walking test is performed while performing a second activity simultaneously. There are many additional task suggestions that can be given during the walk. One of these suggestions is the "counting backwards" task as a cognitive task.
  The test was performed at baseline and after Intervention (8 weeks)
10 Meters Walking Test Under Single Task Condition (10MWTST) | 5 minutes
  Measures the time required to walk 10 meters. Administration time is usually less than 5 minutes. Performed using a "flying start": the patient walks 14 meters and the time is measured for the intermediate 10 meters. The individual walks at their preferred walking speed. It is aimed to measure walking speed.
  The test was performed at baseline and after Intervention (8 weeks)
Tinetti Falls Efficacy Scale (FES) | 5 minutes
  A 10-item questionnaire designed confidence in their ability to perform 10 daily tasks without falling as an indicator of how one's fear of falling impacts physical performance. Each item is rated from 1 ("very confident") to 10 ("not confident at all"), and the per item ratings are added to generate a summary.
  The test was performed at baseline and after Intervention (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Yüzlü, PT MSc, Principal Investigator — Darüşşafaka Physical Therapy and Rehabilitation Center; Semra Oğuz, PhD, Study Director — Marmara University; Mine Gülden Polat, Prof PhD, Study Chair — Marmara University
Locations (1):
- Darüşşafaka Physical Therapy and Rehabilitation Center, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuzlu V, Oguz S, Timurtas E, Aykutoglu E, Polat MG. The Effect of 2 Different Dual-Task Balance Training Methods on Balance and Gait in Older Adults: A Randomized Controlled Trial. Phys Ther. 2022 Mar 1;102(3):pzab298. doi: 10.1093/ptj/pzab298. PMID 34972869